CLINICAL TRIAL: NCT05170126
Title: ZEPOSIA® (Ozanimod) Pregnancy Registry: A Prospective, Observational Study on the Safety of Ozanimod Exposure in Pregnant Women and Their Offspring
Brief Title: A Study on the Safety of Ozanimod Exposure in Pregnant Women and Their Offspring
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-003
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Ozanimod; Pregnancy; Outcomes; Obstetric; Infant
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

GROUPS / COHORTS (3):
- Ozanimod-exposed participants: Women with a diagnosis of multiple sclerosis (MS) who are exposed to ozanimod during the exposure window.
- Comparator-exposed participants: Women with a diagnosis of MS who are not exposed to ozanimod or other sphingosine 1-phosphate (S1P) therapies during the exposure window but who are exposed to other products approved to treat MS during the exposure window.
- Unexposed participants: Women with a diagnosis of MS who are not exposed to ozanimod or other products approved to treat MS during the exposure window.

SUMMARY:
The purpose of this study is to provide information on maternal, fetal, and infant outcomes following exposure of ozanimod during pregnancy so that participants and physicians can weigh the benefits and risks of exposure to the pharmaceutical during pregnancy and make informed treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple sclerosis (MS)
* Currently or recently pregnant
* Reside in the United States, Canada or Germany.

Exclusion Criteria:

• Exposure to other S1P therapies, cladribine, or mitoxantrone during the first trimester.

Other protocol-defined inclusion/exclusion criteria apply

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: The study population will include pregnant women of any age who reside in the United States, Canada or Germany.
Sampling Method: Probability Sample
Enrollment: 1182 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformations | Up to first year of life

SECONDARY OUTCOMES:
Minor congenital malformations | Up to first year of life
Pre-eclampsia | Through pregnancy
Eclampsia | Through pregnancy
Spontaneous abortion | Through pregnancy
Stillbirth | Through pregnancy
Elective termination | Through pregnancy
Preterm birth | Through pregnancy
Small for gestational age | Up to first year of life
Postnatal growth deficiency | Up to first year of life
Infant developmental deficiency | Up to first year of life
Perinatal death | Up to first year of life
Neonatal death | Up to first year of life
Infant death | Up to first year of life
Serious or opportunistic infant infection (SOI) | Up to first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (2):
  - Evidera INC., Bethesda, Maryland
  - Evidera, Bethesda, Maryland
- Marienhospital Herne, Klinikum Der Ruhr-Universitaet Bochum, Herne, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html